CLINICAL TRIAL: NCT06896266
Title: Understanding and Characterizing the Genetics of Patients With Arrhythmia-Induced Cardiomyopathy
Brief Title: Genetic Characterization of Patients With Arrhythmia-Induced Cardiomyopathy
Acronym: UNCHAINED-I
Status: Recruiting | Type: Observational
Sponsor: Hospital Universitario 12 de Octubre (Other)
Responsible Party: Principal Investigator, Martín Negreira-Caamaño, MD, PhD, MD, PhD, Hospital Universitario 12 de Octubre
Other Study IDs: 24/391
Record Dates: First submitted 2025-03-13; First posted 2025-03-26 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Arrhythmia; Cardiomyopathy; Arrhythmia-induced Cardiomyopathy (AiCM)
Keywords: atrial fibrillation; atrial flutter; heart failure; arrhythmia-induced cardiomyopathy; cardiomyopathy; genetics
MeSH Terms: conditions — Arrhythmias, Cardiac; Cardiomyopathies; Atrial Fibrillation; Atrial Flutter; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- A: Patients with arrhytmia-induced cardiomyopathy criteria
- B: Patients without arrhytmia-induced cardiomyopathy criteria

SUMMARY:
The goal of this observational study is to learn about the genetic insights of arrhythmya-induced cardiomyopathy and its clinical prognosis. The main questions it aims to answer are:

I. Does patients with arrhythmia-induced cardiomyopathy have a greater proportion of genetic mutations compared with other types of cardiomyopathy or general population? II. Have the genetics any prognostic impact in patients with arrhythmia-induced cardiomyopathy?

DETAILED DESCRIPTION:
This is a multicentric prospective observational study including patients with suspected arrhythmia-induced cardiomyopathy (AiC) and undergoing rhythm control strategy. AiC suspicion is defined by the presence of left ventricular ejection fraction <50% with no other more plausible explanation than a new-onset arrhythmia.

Patients who met the inclusion/exclusion criteria will be followed during 1 year after the rhythm control procedure (electric cardioversion or catheter ablation) to asess rhythm control status, imaging remodeling and clinical events. A genetic test will be performed during the study time to asess the existace of genetic variants in cardiomyopathy-related genes. Follow-up visits will be scheduled at 2, 6 and 12 months after inclusion and electrocardiogram and echocardiography will be performed.

AiC will be confirmed in case of left ventricular ejection fraction recovery >10% or absolute value >54% during the follow up imaging evaluations.

Primary analysis will asess the prevalence of pathogenic /likely patogenic variants in patients fullfilling AiC criteria and compared with those who not (without AiC). Secondary analysis will be focused on the incidence of cardiovascular events (heart failure-related and rhythm control-related) during the follow up and its relationship with the genetic background and the AiC status.

Imaging test during follow up will be performed and changes in ventricular and atrial parameters will be used to asess cardiac remodeling.

Further rhythm control asessment will be performed following routinary clinical practice in each participant center.

ELIGIBILITY:
Inclusion Criteria:

* Presence of atrial fibrillation or atrial flutter not self-limited.
* Performance of a cardiac imaging test with systolic function analysis (echocardiogram, magnetic resonance, CT scan) during the clinical course of the arrhythmia, exhibiting a left ventricular ejection fraction (LVEF) <50%. In order for the test to be representative, the maximum time between the performance of the imaging test and the rhythm control procedure will be 3 months, in the absence of intervening cardiovascular events that may have caused a variation in LVEF. In the event that the patient had a previously known LVEF <50%, the change with respect to this attributable to tachyarrhythmia has to be ≥10%.
* Signature of informed consent.
* Ability to understand and accept participation in the study.

Exclusion Criteria:

* Refusal of informed consent.
* Legal or juridical incapacity.
* Age <18 years.
* Life expectancy less than 1 year.
* Impossibility of a follow-up of at least 6 months.
* Presence of a ventricular rate >140 beats per minute, limiting the validity of imaging measurements.
* Presence of known factors causing systolic ventricular dysfunction:

  * Prior cardiomyopathy diagnosis.
  * Severe mitral or aortic valve disease.
  * Non-revascularizable ischemic heart disease.
  * Context of peri-resuscitation cardiopulmonary care.
  * Abusive alcohol consumption, defined as >80 grams of ethanol or >7 standard alcoholic beverages per day.
  * Active treatment with chemotherapeutic agents or radiation therapy to the thorax.
  * Known infection with Trypanosoma cruzi, Borrellia burgdorferi or other infectious agent causing cardiomyopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with clinical suspected arrhythmia-induced cardiomyopathy
Sampling Method: Non-Probability Sample
Enrollment: 109 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of pathogenic or likely pathogenic variants in genetic test | Through study completion, an average of 1 year
  Presence of pathogenic/likely pathogenic genetic variant in genetic test

SECONDARY OUTCOMES:
Heart Failure Admission | Through study completion, an average of 1 year
  Incidence of new hospitalización or urgent visit due to heart failure requiring intravenous diuretics
Arrhythmia recurrence | Through study completion, an average of 1 year
  Incidence of any atrial tachyarrhytmia (Atrial fibrillation, atrial flutter or atrial tachycardia) conditioning an atrial rate >150 beats per minute and with a duration of >5 minutes.
New unplanned rhythm control procedure | Through study completion, an average of 1 year
  Incidence of unplanned electrical cardioversion or catheter ablation of an atrial tachyarrhythmia (Atrial fibrillation, atrial flutter or atrial tachycardia)
Atrial reverse remodelling | Through study completion, an average of 1 year
  Incidence of atrial reverse remodelling (ARR). ARR will be considered with a decrease in >1 degree of atrial dilatation (0=non dilated; 1= mild; 2=moderate; 3=severe) or a decrease >15% in the left atrial indexed volume

OTHER OUTCOMES:
Cardiovascular Hospitalization | Through study completion, an average of 1 year
  Incidence of unplanned hospital admission due to a cardiovascular aethiology, including acute coronary syndrome, rhythm disorder, heart failure, valvular heart disease, cardiogenic syncope, ischaemic stroke or transient ischaemic attack, acute aortic syndrome, pulmonary or systemic embolism or unexplained sudden cardiac death.
Mortality | Through study completion, an average of 1 year
  Death of any cause. Cardiovascular death will be also asesed

CONTACTS AND LOCATIONS:
Overall Officials: Martín Negreira-Caamaño, MD, PhD, Study Director — Cardiology department, 12 de Octubre University Hospital; Rafael Salguero-Bodes, MD, Study Director — Cardiology Department, 12 de Octubre University Hospital
Locations (4):
- Spain (4):
  - Ciudad Real General University Hospital, Ciudad Real, Castille-La Mancha
  - 12 de Octubre University Hospital, Madrid, Madrid
  - Albacete University Hospital Complex, Albacete
  - Ramón y Cajal University Hospital, Madrid

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Serban T, Badertscher P, du Fay de Lavallaz J, Providencia R, Migliore F, Mugnai G, Penela D, Perrotta L, Kuhne M, Sticherling C, Chun KJ. Definition and management of arrhythmia-induced cardiomyopathy: findings from the European Heart Rhythm Association survey. Europace. 2024 May 2;26(5):euae112. doi: 10.1093/europace/euae112. PMID 38693772
- [Background] Shoureshi P, Tan AY, Koneru J, Ellenbogen KA, Kaszala K, Huizar JF. Arrhythmia-Induced Cardiomyopathy: JACC State-of-the-Art Review. J Am Coll Cardiol. 2024 Jun 4;83(22):2214-2232. doi: 10.1016/j.jacc.2024.03.416. PMID 38811098